CLINICAL TRIAL: NCT01763736
Title: Medical Use of Song In Critical Care (MUSIC)
Acronym: MUSIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Gerald L. Weinhouse, Physician, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012-P-002287
Record Dates: First submitted 2013-01-03; First posted 2013-01-09 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Stress; Anxiety; Sleep
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Music (Experimental): Everyone enrolled with receive music sessions.
  Interventions: Behavioral: Music

INTERVENTIONS:
Behavioral: Music — playlist per patient preference

SUMMARY:
The objective of this research study is to assess the effects of music on patients' experience in the Intensive Care Unit (ICU). The hypothesis of this study is that patients who receive music therapy will report a reduction in negative recollections and experiences while on mechanical ventilation and will require fewer pharmacologic agents to maintain their sedation.

DETAILED DESCRIPTION:
Music therapy has been applied in a variety of clinical settings to reduce stress, provide a distraction for patients from unpleasant procedures or symptoms, and improve the overall atmosphere and general comfort of patients.

In a preliminary study, investigators have found that subjects experience symptoms of anxiety and stress. It is the investigators hope that providing music as an intervention will alter subjects' recollections of their time in the ICU and creates a more positive ICU experience.

The investigator aims to provide the music intervention, receive full questionnaire completion and recall of subjects' experiences from a total of 40 subjects. Some subjects, however, will not have recall of either the ICU or mechanical ventilation and, therefore, it is predicted that it will require enrolling approximately 75 subjects to reach this goal.

The music intervention will begin after surrogate consent is obtained. Each day while mechanically ventilated, the subject will receive a morning and an afternoon music session lasting one hour. If available, single subject use, disposable headphones may be utilized, or music may be played directly through the computer speakers. Music sessions will occur each day while the subject is mechanically ventilated or up to seven consecutive days. During each music session, study staff will complete a clinical assessment(consisting of vital signs, ventilation data and medications) at three time points during each music session. It is anticipated that some subjects may only have 1 music session per day, or have to skip a day due to clinical condition. If a subject is only able to have one music session on a specific day or a day is missed, a subject will not be considered withdrawn from the study or ineligible for further participation. This will be recorded on the source documents, and the total number of music sessions will be analyzed during analysis. In addition, study staff will not preclude additional music sessions if requested by surrogates. This will also be documented in the source documents by study staff.

Subjects that receive any music sessions during mechanical ventilation will be approached after their discharge from the ICU and before discharge from the hospital. At this point in the study, subjects will be asked to sign the consent form themselves, indicating that they agree to continue with the study and complete the questionnaires. The Mini Mental Status Exam will be done to assess capacity to complete the ICU Stressful Experiences Questionnaire. A score of 25 or higher will be used as a marker to determine if a subject will be administered the questionnaire as was done in the prior study. If potential candidates are deemed to have capacity they will be administered the 32-item, previously validated, ICU Stressful Experiences Questionnaire with the addition of a few questions specific to their recall and experience with the music while critically ill. If a subject receives music sessions, but is not able to provide consent for the questionnaires (due to clinical limitations or hospital discharge) they will not be excluded from the study. A limited data set will be utilized for these subjects.

After the questionnaire has been administered, medical record data will be abstracted from the chart.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 yrs of age
* Admitted to Medical Intensive Care Unit (MICU) (3B and 3C) or Surgical Intensive Care Unit (SICU) (8C, 8D, 11C)
* Expected to receive mechanical ventilation ≥ 24hr
* Surrogate present to provide informed consent

Exclusion Criteria:

* Intubated at a transferring hospital for > 24 hr before arrival to Brigham and Women's Hospital (BWH)
* Chronically ventilator dependent before admission to the hospital
* Transplant candidate or recipient
* Non-English speaking as the questionnaire has not been translated
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Response on ICU Stressful Experiences Questionnaire | After discharge from the ICU, while still in hospital (expected 5-10 days after hospital admission)
  A 32-item, previously validated, ICU Stressful Experiences Questionnaire with the addition of a few questions specific to their recall and experience with the music while critically ill will be administered. Responses will be used to determined subject recall of the ICU and music intervention.

SECONDARY OUTCOMES:
Change in vital signs | Pre-music intervention and during music intervention
  Vital signs will be recorded before and during each music session. (Heart rate, blood pressure, respiratory rate, oxygen saturation, etc.)Vital signs before music session will be compared to vital signs during music session to look for any significant changes.
Change in Vital Signs | Before music intervention and after intervention
  Vital signs will be recorded before and after each music session. (Heart rate, blood pressure, respiratory rate, oxygen saturation, etc.)Vital signs before music session will be compared to vital signs aftermusic session to look for any significant changes.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Weinhouse, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States